CLINICAL TRIAL: NCT02736344
Title: BioNIR Ridaforolimus Eluting Coronary Stent System (BioNIR) In Coronary Stenosis - PK Study
Brief Title: BIONICS - Pharmacokinetics (PK) Trial
Acronym: BIONICS
Status: Completed | Type: Observational
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BioNIR PK- 001
Record Dates: First submitted 2016-03-15; First posted 2016-04-13 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2021-08

CONDITIONS: Heart Disease
Keywords: coronary luminal diameter; lesions; vessels
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BioNIR Ridaforolimus (drug eluting stent (DES): The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0
  The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
  Interventions: Device: BioNIR Ridaforolimus Eluting Coronary Stent

INTERVENTIONS:
Device: BioNIR Ridaforolimus Eluting Coronary Stent

SUMMARY:
The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:

* Stent - mounted Cobalt Chromium (CoCr) alloy based stent
* Delivery System - Rapid Exchange (RX) Coronary System
* Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and polymer coating (CarboSil®)
* Ridaforolimus drug - Chemical Abstracts Service (CAS) Registry Number: 572924-54-0 The product is indicated for improving coronary luminal diameter in patients with symptomatic heart disease due to lesions in vessels with reference diameters of 2.5mm to 4.25mm, including complex lesions.

DETAILED DESCRIPTION:
The study will be a prospective, multicenter, single-arm study involving up to 4 centers in the US.

The subject population is subjects with an indication for percutaneous coronary intervention (PCI) with stent implantation for stable angina and/or silent ischemia. Twelve (12) consecutive patients referred for PCI or possible PCI with suspected or proven coronary artery disease will be screened and consented.

Twelve (12) consecutive patients referred for PCI or possible PCI with suspected or proven coronary artery disease will be screened and consented. Patients with ACS are not eligible. Patients will be considered enrolled and eligible to receive the BioNIR stent after successful and uncomplicated crossing of the target lesion and successful and uncomplicated lesion preparation (such as pre-dilatation) if needed. At least 30% (4 subjects) will receive more than one stent or a sufficiently long stent so that the total implanted stent dose is >1.5 times the ridaforolimus dose of the workhorse BioNIR stent (3.0x17 mm).

For each patient, a total of up to 14 blood samples will be collected at the following time points: immediately prior to the first stent implant as time 0, at 10 and 30 minutes, and at 1, 2, 4, 8, 12, 24±6, 48±12, 72±12, 168±36 (7 days), 336±36 (14 days) and 720±36 hours (30 days) after the first BioNIR stent implantation. Whole blood concentration of ridaforolimus will be determined using a validated high performance liquid chromatography mass spectrometry/mass spectrometry (HPLC-MS/MS) method. If two consecutive measurements are available and both demonstrate ridaforolimus levels below the detection limit of the assay, the levels at all subsequent time points will not need to be measured.

Relationship to BIONICS STUDY: The general and angiographic inclusion and exclusion criteria will be identical to the pivotal BIONICS trial with the exception of Acute Coronary Syndrome (ACS) patients who will be excluded. Clinical data will be collected in an identical manner to the BIONICS study.

(Clinical follow-up will be performed at 30 days, 6 months, and 1, 2, 3, 4, and 5 years post enrollment.) The following pharmacokinetic parameters will be evaluated: maximum concentration (Cmax), Cmax adjusted by treatment dose, time to maximum concentration (tmax), the time of the last quantifiable concentration (tlast ), half-life time ( t1/2), total area under the concentration-time curve from time 0 to tlast (AUC0-tlast), total area under the concentration-time curve from time 0 to tlast (AUC0-t∞) and total body clearance (CL). AUCs normalized by treatment dose will also be derived.

12 subjects will be enrolled in order to evaluate the pharmacokinetic parameters of ridaforolimus release from the BioNIR stent. The number of subjects was chosen based on experience in the literature from other 'limus' drug eluting stents as well as specific request from FDA.

ELIGIBILITY:
General Inclusion:

1. Stable patients (non-ACS) with an indication for possible PCI for stable angina, and/or silent ischemia (in absence of symptoms a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or Fractional Flow Reserve (FFR) ≤0.80 must be present).
2. Patient is willing and able to provide informed written consent and comply with follow-up visits and testing schedule

Angiographic Inclusion Criteria:

1. Target lesion(s) must be located in a native coronary artery or bypass graft conduit with visually estimated diameter of ≥2.5mm to ≤4.25mm
2. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus that is non-occlusive and does not require thrombectomy, chronic total occlusion (CTO), bifurcation lesions (except planned dual stent implantation), ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions, and saphenous vein graft lesions.
3. Overlapping stents are allowed

General Exclusion Criteria:

1. PCI with previous BioNIR stent implantation.
2. ACS within 1 month of enrollment.
3. Patients receive strong CYP3A inhibitors or inducers such as Ketoconazole or Rifampin.
4. PCI within the 24 hours preceding the baseline procedure.
5. Non-target lesion PCI in the target vessel within 12 months of the baseline procedure.
6. History of stent thrombosis.
7. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including intra aortic balloon pumping (IABP).
8. Subject is intubated.
9. Known left ventricular ejection fraction (LVEF) <30%.
10. Relative or absolute contraindication to duale antiplatelet therapy (DAPT) for 12 months (including planned surgeries that cannot be delayed)
11. Subject has an indication for chronic oral anticoagulant treatment (with either vitamin K antagonists or novel anticoagulants (NOACs)
12. Calculated creatinine clearance <30 mL/min using Cockcroft-Gault equation.
13. Hemoglobin <10 g/dL.
14. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
15. White blood cell (WBC) count <3,000 cells/mm3.
16. Clinically significant liver disease.
17. Active peptic ulcer or active bleeding from any site.
18. Bleeding from any site within the prior 8 weeks requiring active medical or surgical attention.
19. If femoral access is planned, significant peripheral arterial disease which precludes safe insertion of a 6French (6F) sheath.
20. History of bleeding diathesis/coagulopathy/will refuse blood transfusions.
21. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attributed to cerebrovascular accident (CVA).
22. Known allergy to the study stent components, e.g. cobalt, nickel, chromium, molybdenum, Carbosil®, PBMA, Biolinx polymer, or limus drugs (ridaforolimus, zotarolimus, tacrolimus, sirolimus, everolimus, or similar drugs or any other analogue or derivative or similar compounds).
23. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
24. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease).
25. Patient participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
26. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within 1week before treatment).
27. Women who intend to become pregnant within 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
28. Patient has received / is on a waiting list for an organ transplant.
29. Patient is receiving or scheduled to receive chemotherapy within 30 days before or any time after the baseline procedure.
30. Patient is receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive disease (e.g., HIV). Corticosteroids are allowed

    Angiographic exclusion criteria:
31. Target lesions in more than two (2) major coronary arteries (ie, two of left anterior descending artery [LAD], LCX, RCA) including their respective branches (the Ramus Intermedius is defined as a branch of the LCX).
32. More than two target lesions per target vessel are planned (two lesions separated by less than 10 mm that can be covered by a single stent are considered as one lesion).
33. More than 100mm length planned study stenting in entire coronary tree.
34. Occlusive thrombus and/or thrombus requiring thrombectomy in a target vessel.
35. Unprotected left main lesions ≥30%, or planned unprotected left main intervention.
36. Ostial LAD or LCX target lesions (stenting of any diseased segment within 5 mm of the unprotected left main coronary artery).
37. Target Bifurcation lesions with planned dual stent implantation.
38. Stenting of target lesions due to DES restenosis.
39. Another lesion in a target or non-target vessel (including all side branches) is present that requires or has a high probability of requiring PCI within 12 months after the baseline procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an indication for percutaneous coronary intervention (PCI) with stent implantation for stable angina and/or silent ischemia.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | For each patient, a total of up to 14 blood samples will be collected at the following time points: immediately prior to the first stent implant as time 0, at 10 and 30 minutes, and at 1, 2, 4, 8, 12, 24±6, 48±12, 72±12, 168±36 hours.
  Maximum concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizik, MD, Principal Investigator — Scottsdale Heart Group
Locations (2):
- United States (2):
  - Scottsdale Heart Group, Scottsdale, Arizona
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan

IPD SHARING:
Plan to Share IPD: No